CLINICAL TRIAL: NCT01459744
Title: An Intervention to Improve ICD Deactivation Conversations (WISDOM - Working to Improve discuSsions About DefibrillatOr Management)
Brief Title: An Intervention to Improve Implantable Cardioverter-Defibrillator Deactivation Conversations
Acronym: WISDOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Colorado, Denver (Other); Mayo Clinic (Other); University of Pennsylvania (Other); Oregon Health and Science University (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GCO 09-0618; 1R01HL102084-01A1 (NIH)
Record Dates: First submitted 2011-10-13; First posted 2011-10-26 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Communication; Heart Failure
Keywords: Heart failure; Palliative care; Communication
MeSH Terms: conditions — Communication; Heart Failure | interventions — Cardiologists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Communication training for cardiologists (Experimental): The intervention consists of an educational workshop for heart failure physicians, a reminder system, and a system providing aggregated feedback on their conversations with patients about ICD deactivation.
  Interventions: Behavioral: Communication training for cardiologists.
- Control arm (Placebo Comparator): Cardiology grand rounds will be held at usual care sites on the importance of advance care planning.
  Interventions: Other: Control arm

INTERVENTIONS:
Behavioral: Communication training for cardiologists. — Communication training: a 90 minute workshop to discuss ways to improve communication in patients with serious illness.
  Reminders to Cardiologists. Cardiologists will receive reminders to prompt them to have conversations relating to ICD management with patients enrolled in the study.
  Audit and feedback. Cardiologists will receive feedback on their rates of conversation as well as data on patient/family satisfaction with their communication skills.
  Arms: Communication training for cardiologists
Other: Control arm — Cardiology grand rounds will be held at usual care sites on the importance of advance care planning.
  Arms: Control arm

SUMMARY:
An Implantable Cardioverter-Defibrillator (ICD) is a device implanted in a patient's chest to monitor the heart rhythm and deliver shocks to terminate potentially lethal arrhythmias when necessary. While ICDs reduce sudden cardiac death, patients with ICDs eventually die of heart failure or other diseases. As patients near the end of life, physiologic changes (intrinsic and extrinsic to the heart) may affect the cardiac conduction system, leading to more arrhythmias and increasing the frequency of shocks. Because ICD shocks can cause pain and anxiety and may not prolong a life of acceptable quality, it is appropriate to consider deactivating the shocking function of ICDs as patients' clinical status worsens and death is near. This will be a randomized controlled trial of a physician centered counseling and education intervention to improve clinician-patient communication about the management of ICDs.

DETAILED DESCRIPTION:
An Implantable Cardioverter-Defibrillator (ICD) is a device implanted in a patient's chest to monitor the heart rhythm and deliver shocks to terminate potentially lethal arrhythmias when necessary. While ICDs reduce sudden cardiac death, patients with these devices do eventually die, either of heart failure or other chronic diseases. As a patient's disease worsens, physiologic changes (intrinsic and extrinsic to the heart) may affect the cardiac conduction system, leading to more arrhythmias and increasing the frequency of shocks. Because ICD shocks can cause pain and anxiety and may not prolong a life of acceptable quality, it is appropriate to consider ICD deactivation as a patient's clinical status worsens and death is near. However, these conversations rarely occur. The investigators propose to conduct a randomized clinical trial of a physician-centered patient counseling and support intervention to improve communication between cardiologists and patients with ICDs. The goals of the study are to determine the effectiveness of the intervention to: 1) increase conversations about ICD deactivation, 2) increase the number of patients who have their devices deactivated, and 3) improve mental health outcomes for bereaved caregivers of deceased patients. The unit of randomization is the hospital, the intervention is aimed at cardiologists, and the unit of analysis is the patient. The investigators have created a network of six academic medical centers across the country. The intervention to be delivered consists of three parts. First, the PI will conduct a workshop on communication specific to ICD-deactivation with cardiologists at the intervention centers. Second, when enrolled patients are admitted to the hospital or seen in the outpatient setting, the cardiologist will receive two reminders (one via email, one in the patient chart) that the patient is appropriate for a conversation about ICD deactivation. Finally, cardiologists will receive aggregated feedback about the number of conversations they have conducted and data on patients' satisfaction with conversations every six months. Physicians at usual care hospitals receive a didactic lecture on advance care planning. All patients and surrogates will be interviewed at baseline and then assessed at regular intervals to determine the outcomes of: 1) the prevalence of conversations about ICD deactivation as reported by the patient/surrogate; and 2) the frequency with which patients have their devices deactivated. Caregivers will continue to be interviewed at regular intervals up to 6 months after the patient dies to determine the relationship of the intervention to caregiver mental health outcomes. Given the exponential increase in the number of patients with ICDs, this intervention has the potential to improve the quality of care for thousands of patients near the end of life and their families.

ELIGIBILITY:
Inclusion Criteria:

Clinicians:

* At all sites, a core group of approximately 10 heart failure clinicians (physicians, nurses) care exclusively for patients with advanced heart failure in both inpatient and outpatient settings; all of these clinicians are eligible..

Patients:

* Patient does not currently have a ventricular assist device
* Age > 18
* Fluent in English
* Consistent and reliable access to a phone

For Inpatient:

* Has had at least 1 other heart failure in the last year, OR
* Meets all three of the following criteria at time of admission:

  1. BUN > 43
  2. SBP ≤ 115
  3. CR > 2.75 OR
* Was on inotropes OR intravenous diuretics OR intravenous heart failure treatments in emergency department OR in outpatient setting prior to the current hospital admission

For Outpatient

* Has had 2 or more heart failure related admissions in the last year OR
* Has class IV heart failure in the outpatient setting OR
* Has Class III heart failure in outpatient setting AND 1 heart failure related admission in the last year OR
* Has Class III heart failure in outpatient setting AND 2 of the following 4 conditions:

  1. Age ≥ 70
  2. BUN ≥ 43
  3. Cr ≥ 2.75
  4. SBP≤115 OR
* Is on inotropes (e.g., dobutamine, milrinone) OR intravenous diuretics OR intravenous heart failure treatments in emergency department OR in outpatient setting

Caregivers:

* Age > 18
* Fluent in English
* Consistent and reliable access to a phone

Exclusion Criteria for patients:

* Not having an ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of Conversations about ICD Deactivation | after 1st clinical encounter after enrollment for intervention group
  Whether deactivation discussion occurred difference between 1st and 3rd clinical encounters after enrollment
Prevalence of Conversations about ICD Deactivation | 3rd clinical encounter after enrollment for intervention group
  Whether deactivation discussion occurred difference between 1st and 3rd clinical encounters after enrollment
Prevalence of Conversations about ICD Deactivation | 3 months after enrollment for control group
  Whether deactivation discussion occurred difference between 3 and 9 months after enrollment
Prevalence of Conversations about ICD Deactivation | 9 months after enrollment for control group
  Whether deactivation discussion occurred difference between 3 and 9 months after enrollment

SECONDARY OUTCOMES:
Prevalence of ICD Deactivation | After 1st encounter after enrollment for intervention group
  Whether ICD deactivation occurred difference between 1st and 3rd clinical encounters after enrollment
Prevalence of ICD Deactivation | After 3rd encounter after enrollment for intervention group
  Whether ICD deactivation occurred difference between 1st and 3rd clinical encounters after enrollment
Prevalence of ICD Deactivation | After 3 months after enrollment for control group
  Whether ICD deactivation occurred difference between 3 and 9 months after enrollment
Prevalence of ICD Deactivation | After 6 months after enrollment for control group
  Whether ICD deactivation occurred difference between 3 and 9 months after enrollment
Psychological Outcomes in Bereaved Caregivers | 4 weeks after patient death
Psychological Outcomes in Bereaved Caregivers | 6 months after patient death

CONTACTS AND LOCATIONS:
Overall Officials: Nathan E. Goldstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - University of Colorado - Denver, Denver, Colorado
  - Yale New-Haven Hospital, New Haven, Connecticut
  - Mayo Medical Center, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Buxton AE, Lee KL, Fisher JD, Josephson ME, Prystowsky EN, Hafley G. A randomized study of the prevention of sudden death in patients with coronary artery disease. Multicenter Unsustained Tachycardia Trial Investigators. N Engl J Med. 1999 Dec 16;341(25):1882-90. doi: 10.1056/NEJM199912163412503. PMID 10601507
- [Background] Moss AJ, Hall WJ, Cannom DS, Daubert JP, Higgins SL, Klein H, Levine JH, Saksena S, Waldo AL, Wilber D, Brown MW, Heo M. Improved survival with an implanted defibrillator in patients with coronary disease at high risk for ventricular arrhythmia. Multicenter Automatic Defibrillator Implantation Trial Investigators. N Engl J Med. 1996 Dec 26;335(26):1933-40. doi: 10.1056/NEJM199612263352601. PMID 8960472
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Glikson M, Friedman PA. The implantable cardioverter defibrillator. Lancet. 2001 Apr 7;357(9262):1107-17. doi: 10.1016/S0140-6736(00)04263-X. PMID 11297981
- [Background] Eckert M, Jones T. How does an implantable cardioverter defibrillator (ICD) affect the lives of patients and their families? Int J Nurs Pract. 2002 Jun;8(3):152-7. doi: 10.1046/j.1440-172x.2002.00357.x. PMID 12000634
- [Background] Sears SF Jr, Conti JB. Quality of life and psychological functioning of icd patients. Heart. 2002 May;87(5):488-93. doi: 10.1136/heart.87.5.488. No abstract available. PMID 11997430
- [Derived] Gelfman LP, Sudore RL, Mather H, McKendrick K, Hutchinson MD, Lampert RJ, Lipman HI, Matlock DD, Swetz KM, Pinney SP, Morrison RS, Goldstein NE. Prognostic Awareness and Goals of Care Discussions Among Patients With Advanced Heart Failure. Circ Heart Fail. 2020 Sep;13(9):e006502. doi: 10.1161/CIRCHEARTFAILURE.119.006502. Epub 2020 Sep 2. PMID 32873058
- [Derived] Goldstein NE, Mather H, McKendrick K, Gelfman LP, Hutchinson MD, Lampert R, Lipman HI, Matlock DD, Strand JJ, Swetz KM, Kalman J, Kutner JS, Pinney S, Morrison RS. Improving Communication in Heart Failure Patient Care. J Am Coll Cardiol. 2019 Oct 1;74(13):1682-1692. doi: 10.1016/j.jacc.2019.07.058. PMID 31558252